CLINICAL TRIAL: NCT02750397
Title: Prospective Study of HIV+ Deceased Donor Transplant for HIV+ Recipients
Brief Title: HIV-to-HIV Transplant at MGH
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Nahel Elias, M.D., Surgical Director, Kidney Transplant, Massachusetts General Hospital
Other Study IDs: 2016P000355
Record Dates: First submitted 2016-04-21; First posted 2016-04-25 (Estimated); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: HIV; Awaiting Organ Transplant
Keywords: HIV; Kidney Transplant; Liver Transplant; Transplant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- HIV D+/R+: HIV+ recipients who receive an organ transplant from an HIV+ donor
- HIV D-/R+: HIV+ recipients who receive an organ transplant from an HIV- donor

SUMMARY:
HIV-infected (HIV+) individuals who agree to accept and receive a solid organ transplant from an HIV+ deceased donor will be followed to determine the safety and efficacy of this practice. HIV+ individuals who receive a solid organ transplant from HIV-uninfected donors will also be followed.

DETAILED DESCRIPTION:
This is an observational study designed to evaluate safety and outcomes of solid organ transplantation in HIV+ recipients of HIV+ deceased donors. This study will evaluate overall survival and graft survival compared to transplantation with an HIV- organ.

In addition the study will assess potential complications of organ transplant using HIV+ deceased donors - including but not limited to - HIV superinfection, incidence and severity of graft rejection, recurrence of HIV-associated nephropathy, incidence of bacterial infections, and opportunistic infections.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is able to understand and provide informed consent
2. Participant meets standard listing criteria for transplant.
3. Documented HIV infection (by any licensed ELISA and confirmation by Western Blot, positive HIV ab IFA, or documented history of detectable HIV-1 RNA).
4. Participant is ≥ 18 years old.
5. Opportunistic Complications: None or previous history of protocol allowed opportunistic infections or neoplasms with appropriate acute and maintenance therapy and no evidence of active disease.
6. Participant CD4+ T-cell count is >/= 200/μL prior to renal transplant or for liver transplant is >/= 100/μL within 16 weeks prior to transplant and no history of opportunistic infection (OI); or ≥200 μL if history of OI is present.
7. Participant HIV-1 RNA < 50 copies/mL (by any FDA-approved assay performed in CLIA-approved laboratory), in the 26 weeks prior to transplant. Non-consecutive viral "blips" between 50-400 copies RNA/mL will be allowed.
8. Antiretroviral therapy: To avoid drug interactions, ritonavir or cobicistat-containing regimens are not recommended, unless in the opinion of the HIV/Transplant Infectious Disease team there is no alternative regimen expected to control HIV replication.
9. Participant is willing to use PCP, herpes virus and fungal prophylaxis as indicated.

Exclusion Criteria:

1. Participant has concomitant conditions that, in the judgment of the investigators, would preclude transplantation or immunosuppression.
2. Opportunistic Complication History: Any history of progressive multifocal leukoencephalopathy (PML), chronic intestinal cryptosporidiosis of > 1 month duration, or primary CNS lymphoma.
3. Participant has a history of any neoplasm except for the following: resolved kaposi's sarcoma, in situ anogenital carcinoma, adequatelytreated basal or squamous cell carcinoma of the skin, solid tumors (except primary CNS lymphoma) treated with curative therapy and disease free for more than 5 years. History of renal cell carcinoma requires disease free state for 2 years. History of leukemia and disease-free duration will be per site policy.
4. Participant is pregnant or breastfeeding. Note: Participants who become pregnant post-transplant will continue to be followed in the study and will be managed per clinical practice. Women that become pregnant should not breastfeed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All individuals with end-stage organ disease and HIV infection who meet standard clinical criteria for transplantation and the study inclusion and exclusion criteria will be eligible for participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2016-08; Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-16 (Actual)

PRIMARY OUTCOMES:
Patient Survival | One Year

SECONDARY OUTCOMES:
Graft Survival | One, Two, Three Years
Graft Rejection | One, Two, Three Years
HIV Disease Progression | One, Two, Three Years
Development of antiretroviral resistance and X4 tropic virus | Through study completion, up to three years
Incidence of bacterial, fungal, viral and other opportunistic infections | Through study completion, up to three years
Incidence of other transplant complications (surgical and vascular) | Through study completion, up to three years
Analysis of recurrent HIV associated nephropathy | Through study completion, up to three years
Incidence of post-transplant malignancies | Through study completion, up to three years
Incidence of systemic HIV-superinfection | Through study completion, up to three years
Changes in HIV latent viral reservoir | Through study completion, up to three years

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States